CLINICAL TRIAL: NCT02278367
Title: Clinical Evaluation of 18F-AV-1451
Brief Title: Clinical Evaluation of Flortaucipir F 18
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Avid Radiopharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 18F-AV-1451-A14
Record Dates: First submitted 2014-10-28; First posted 2014-10-30 (Estimated); Results first posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-08

CONDITIONS: Alzheimer's Disease; Traumatic Brain Injury; Depression
MeSH Terms: conditions — Alzheimer Disease; Brain Injuries, Traumatic; Depression | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Flortaucipir PET Scans (Experimental)
  Interventions: Drug: Flortaucipir F18; Procedure: Brain PET scan

INTERVENTIONS:
Drug: Flortaucipir F18 — IV injection, 370 MBq (10 mCi), up to two doses
  Other Names: [F-18]T807; 18F-AV-1451; LY3191748; Tauvid
Procedure: Brain PET scan — positron emission tomography (PET) scan of the brain

SUMMARY:
This study is designed to expand the database of flortaucipir F 18 safety and tau binding as measured by PET imaging and to provide standardized conditions for flortaucipir PET use, data collection and analysis to facilitate companion studies including, but not limited to, longitudinal studies of aging, depression, and traumatic brain injury.

ELIGIBILITY:
Subjects should meet inclusion and exclusion criteria for the companion protocol in addition to the criteria below.

Inclusion Criteria:

* Subjects who have a historical volumetric magnetic resonance imaging (MRI) as part of the companion study

Exclusion Criteria:

* Have clinically significant cardiac, hepatic, renal, pulmonary, metabolic, or endocrine disturbances
* Have a screening electrocardiogram with a corrected QT interval (QTc) > 450 msec if male or QTc > 470 msec if female
* Have a history of additional risk factors for Torsades de Pointes (TdP) or are taking drugs known to cause QT-prolongation. Patients with a prolonged QTc interval in the setting of intraventricular conduction block may be enrolled with sponsor approval
* Have a history of drug or alcohol dependence within the last year, or prior prolonged history of dependence unless approved by the sponsor
* Are females of childbearing potential who are not surgically sterile, not refraining from sexual activity or not using reliable methods of contraception
* Have a history of relevant severe drug allergy or hypersensitivity
* Are patients who have received an investigational medication within 30 days prior to the planned imaging session for this study
* Are patients with current clinically significant unstable medical comorbidities
* Are patients who have received a radiopharmaceutical for imaging or therapy within the past 24 hours prior to the imaging session for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2019-06-26 (Actual); Study Completion 2019-06-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Banner Alzheimer's Institute, Phoenix, Arizona
  - Yale University, New Haven, Connecticut
  - Cleveland Clinic Lou Ruvo Center for Brain Health, Las Vegas, Nevada
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Center for Vital Longevity at the University of Texas at Dallas, Dallas, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Cognitively Impaired: Cognitively impaired subjects receiving a flortaucipir PET scan
- Cognitively Normal: Cognitively normal subjects receiving a flortaucipir PET scan
Period: Overall Study
Arm/Group | Cognitively Impaired | Cognitively Normal
Started | 69 | 110
Completed | 59 | 110
Not Completed | 10 | 0
Not completed — Physician Decision | 5 | 0
Not completed — Withdrawal by Subject | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cognitively Impaired | Cognitively Normal | Total
Number analyzed (Participants) | 69 | 110 | 179
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.7 (7.6) | 70.4 (8.18) | 71.3 (8.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 68 | 102
  Male | 35 | 42 | 77
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 10 | 10
  Not Hispanic or Latino | 69 | 100 | 169
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 5 | 5 | 10
  White | 62 | 105 | 167
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 69 | 110 | 179
MMSE [Mean (Standard Deviation); unit: score on a scale] — Mini-mental status exam (MMSE) is a 30-point questionnaire that is used to measure cognitive impairment. Scores range from 0 to 30 with lower scores representing greater levels of cognitive impairment.
  score on a scale | 21 (4.35) | 29.3 (1.06) | 26.1 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Related to Flortaucipir Administration
Description: Frequency of treatment-emergent adverse events considered related to flortaucipir administration by the study investigator. Related events with a frequency > 1.5% are reported.
  (note: all treatment-emergent adverse events, regardless of relatedness designation, are reported in "Adverse Events" section below).
Time Frame: within 48 hours of drug administration
Measure: Count of Participants; unit: Participants
Arm/Group | Cognitively Impaired | Cognitively Normal
Number analyzed (Participants) | 69 | 110
Participants
  Headache | 0 | 3
  Dysgeusia | 0 | 3

2. Primary Outcome: Flortaucipir PET Scan SUVr
Description: Standard Uptake Value Ratio (SUVr) using a weighted cortical average. For SUVr, a value of 1 or lower signifies no flortaucipir activity above background, values greater than 1 signify increasing flortaucipir activity in the brain.
Time Frame: baseline and follow-up scans
Population: Includes only subjects for whom a quantitative image analysis was possible
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio (SUVr)
Arm/Group | Cognitively Impaired | Cognitively Normal
Number analyzed (Participants) | 63 | 107
standardized uptake value ratio (SUVr)
  Baseline SUVr | 1.3983 (0.3641) | 1.004 (0.04871)
  Follow-up Scan SUVr: number analyzed (Participants) | 40 | 0
  Follow-up Scan SUVr | 1.4404 (0.37426) |

ADVERSE EVENTS:
Time Frame: AEs were collected at scan visit and for 48 hours after flortaucipir administration.
Description: AEs defined as occurring or worsening after injection, within 48 hours, at an imaging visit. AEs occurring after administration, but outside that window were not reported, unless considered attributable to study drug. Note: AE results differ from results reported above because this section reports ALL adverse events, regardless of investigator's designation of relatedness.
Arm/Group | Cognitively Impaired | Cognitively Normal
All-Cause Mortality (participants affected / at risk) | 0/69 | 0/110
Serious Adverse Events (participants affected / at risk) | 0/69 | 0/110
Other Adverse Events (participants affected / at risk) | 6/69 | 16/110
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cognitively Impaired (N=69) | Cognitively Normal (N=110)
headache (Nervous system disorders) | 0 (0) | 5 (5)
dysgeusia (Nervous system disorders) | 0 (0) | 3 (3)
dizziness (Nervous system disorders) | 0 (0) | 1 (1)
paraesthesia (Nervous system disorders) | 0 (0) | 1 (1)
injection site pain (General disorders) | 1 (1) | 1 (1)
asthenia (General disorders) | 0 (0) | 1 (1)
feeling abnormal (General disorders) | 0 (0) | 1 (1)
gait abnormal (General disorders) | 0 (0) | 1 (1)
injection site coldness (General disorders) | 0 (0) | 1 (1)
blood pressure increased (Investigations) | 2 (2) | 2 (2)
dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2)
nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
palpitations (Cardiac disorders) | 1 (1) | 0 (0)
nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
procedural headache (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
loss of bladder sensation (Renal and urinary disorders) | 0 (0) | 1 (1)
hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2014-09-05): https://cdn.clinicaltrials.gov/large-docs/67/NCT02278367/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT02278367/SAP_001.pdf